CLINICAL TRIAL: NCT07248098
Title: Investigation of the Effect of Abdominal Hot Water Bag Application on Pain and Bowel Peristalsis in Individuals Diagnosed With Ileus
Brief Title: Abdominal Hot Water Bag Aplication Ileus Care
Acronym: Ileus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Meltem Akbaş, Dr, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 06.09.2024/147; 06.09.2024/147 (Other: Cukurova University)
Record Dates: First submitted 2025-09-17; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Ileus; Nursing Care; Pain
Keywords: ileus; nursing care; pain; water treatment
MeSH Terms: conditions — Ileus; Pain

STUDY DESIGN:
Intervention Model Description: For the experimental group, heat will be applied to the abdominal area for 10 minutes in the morning and 10 minutes in the evening, starting from the first day of the patient's admission to the clinic. The application will continue for 10 minutes each morning and evening until the patient passes their first gas. Consistent with literature, a water bag filled with hot water at 55 ± 2°C will be wrapped with two towels, and the water temperature will be measured with a thermometer capable of measuring liquid temperature. The water bag will be applied to the abdominal area for 10 minutes with the patient in the supine position.
  Patients in the control group will not be subjected to any postoperative intervention other than routine clinical care practices.
Who Masked: Participant
Masking Description: Participant blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): hot water application
  Interventions: Other: hot water application
- control (No Intervention): standart care

INTERVENTIONS:
Other: hot water application — hot water application
  Arms: intervention

SUMMARY:
The role of nurses in the management of ileus is very important as they are part of the multidisciplinary approach. The study aimed to determine the effect of a hot water bag applied to the abdominal region on pain caused by decreased or cessation of intestinal peristalsis in individuals diagnosed with ileus on reducing or relieving pain and restoring intestinal peristalsis.

DETAILED DESCRIPTION:
The study aimed to determine the effect of a hot water bag applied to the abdominal region on pain caused by decreased or cessation of intestinal peristalsis in individuals diagnosed with ileus on reducing or relieving pain and restoring intestinal peristalsis. Data will be evaluated using a literature-based Patient Personal Information Form, Visual Analog Scale, burping, and auscultation of bowel sounds with a stethoscope. Sample calculations were performed using a priori power analysis (t-test) for the intervention and control groups. Accordingly, with an effect size of d=2.06, a 5% error rate (α=0.01), and 99% power (1-β=0.99), the minimum sample size for both groups was calculated as 54. Considering potential losses, the total sample size was increased by 10%, resulting in 30 patients in each group (Experimental Group: 30, Control Group: 30), and a total of 60 patients.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the study,
* No communication or intellectual disabilities,
* Reading and writing skills,
* Diagnosed with brid ileus, as a type of ileus,
* Adult individuals over the age of 18

Exclusion Criteria:

* Leaving the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-11-22 (Estimated); Study Completion 2025-11-25 (Estimated)

PRIMARY OUTCOMES:
Visiual Analog Scale | 30 day
  It is scored from 1 to 10. The lowest score is 0, meaning no pain, and the highest score is 10, meaning unbearable pain. The higher the score, the greater the pain.

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Akbaş, Dr, Principal Investigator — Cukurova University
Locations (1):
- Cukurova University, Adana, Saricam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No